CLINICAL TRIAL: NCT05852665
Title: Ultrasound-guided Resection of Buccal Mucosal Carcinomas - a Multicenter Study
Brief Title: Buccal Cancer Resection Ultrasound Guided
Acronym: BRUG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Rijnstate Hospital (Other); University Medical Center Groningen (Other); Medisch Spectrum Twente (Other); Medical Center Haaglanden (Other); Antoni van Leeuwenhoek Ziekenhuis (Unknown)
Responsible Party: Principal Investigator, Rob Noorlag, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL83714.041.23
Record Dates: First submitted 2023-04-18; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Buccal Mucosa Cancer; Squamous Cell Carcinoma
Keywords: Buccal mucosal carcinoma; Squamous cell carcinoma; Ultrasound; Multicenter
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasound-guided surgery (Experimental)
  Interventions: Device: Ultrasound-guided resection

INTERVENTIONS:
Device: Ultrasound-guided resection — Ultrasound-guided resection of buccal squamous cell carcinomas

SUMMARY:
The aim of this research is to decrease the number of inadequate tumor-free margins, probably resulting in less adjuvant therapy, less local recurrences and better quality of life.

DETAILED DESCRIPTION:
Buccal mucosa cancer is a rare disease. In the Netherlands, approximately 100 patients are treated for this disease each year. To obtain good local control, it is important that the histological distance from the tumor to the resection plane is 5 mm or more (tumor-free margin). If the tumor-free margin is smaller, such as close (1-5 mm) or involved (<1 mm) margins, there is usually an indication for adjuvant therapy. Now, the tumor-free margins in buccal mucosa cancer are often insufficient, so that a significant proportion of patients require adjuvant treatment (re-resection or radiotherapy). Postoperative radiotherapy can greatly reduce the quality of life due to the development of, for example, osteoradionecrosis, mucositis and fibrosis. During a re-resection it is often difficult to find the location of the insufficient margin. Ultrasound-guided resection can be used to visualize the tumor during surgery, in order to improve the tumor-free margins. Currently, the tumor-free margin is only estimated palpably and frozen sections are sometimes used in case of doubt.

The aim of this research is to decrease the number of involved margins, probably resulting in less adjuvant therapy, less local recurrences, and better quality of life.

In this trial, 50 patients with a squamous cell carcinoma of the buccal mucosa will be included for treatment with ultrasound-guided resection.

50 patients with a squamous cell carcinoma of the buccal mucosa, who will be treated with surgery under general anesthesia, will be included in this study. The tumor has to be visible as an hypo-echogenic region on the ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* buccal mucosal squamous cell carcinoma
* surgical removal under general anesthesia

Exclusion Criteria:

* tumor is not visible on ultrasound as echolucent region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of involved margins | within 2 weeks after surgery
  Number of involved margins

SECONDARY OUTCOMES:
Sensitivity and specificity of ultrasound for identifying involved margins | within 2 weeks after surgery
  accuracy of ultrasound
Number of patients with an indication for local adjuvant therapy | within one month after surgery
  need for local adjuvant treatment
Quality of life assessed by questionnaires at 4 timepoints | before surgery, at 4, 8, and 12 months after surgery
  Influence of treatment on quality of life

IPD SHARING:
Plan to Share IPD: No